CLINICAL TRIAL: NCT07053072
Title: A Prospective，Single Arm Clinicial Trial Evaluating PD-1 mRNA LNP Vaccine for the Treatment of Advanced Primary Hepatocellular Carcinoma Failing Standard Therapy
Brief Title: PD-1 mRNA LNP Vaccine for Advanced Primary Hepatocellular Carcinoma.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD，professor, West China Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-755
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: This single-centre, open-label, single-arm trial uses a dose-escalation framework to evaluate the safety and biological activity of PD-1 mRNA LNP in the treatment of patients with advanced hepatocellular carcinoma who have failed standard therapy. All participants will maintain a fixed chemotherapy/immunotherapy regimen based on their respective malignancies, with only the dose of PD-1 mRNA LNP changing.
  Three cases will be enrolled in each dose group, with the planned dose groups being the 50 μg, 75 μg and 100 μg groups. It consisted of 5 doses of basal immunisation and subsequent personalised treatment. For the base immunisation, the first 4 doses were administered 1 week apart each and the 5th dose was administered 1 month after the 4th dose.
  Dose-limiting toxicity (DLT) will be monitored through a 21-day monitoring window. Escalation decisions will be made using a Bayesian Optimal Interval (BOIN) approach, with DLT classification following the
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): Low-dose PD-1 mRNA LNP vaccine for advanced primary hepatocellular carcinoma failing standard therapy
  Interventions: Drug: Low Dose PD-1 mRNA LNP Vaccine
- Medium Dose (Experimental): Medium Dose PD-1 mRNA LNP Vaccine for Advanced Primary Hepatocellular Carcinoma Failing Standard Treatment
  Interventions: Drug: Medium dose PD-1 mRNA LNP vaccines
- High Dose (Experimental): High Dose PD-1 mRNA LNP Vaccine for Advanced Primary Hepatocellular Carcinoma Failing Standard Treatment
  Interventions: Drug: High dose PD-1 mRNA LNP vaccines

INTERVENTIONS:
Drug: Low Dose PD-1 mRNA LNP Vaccine — Patients will receive PD-1 mRNA LNP vaccine at 50 mcg weekly for the first 4 doses and a 5th dose 1 month after the 4th dose.
  Other Names: PD-1 mRNA LNP vaccine at 50 mcg
  Arms: Low Dose
Drug: Medium dose PD-1 mRNA LNP vaccines — Patients will receive PD-1 mRNA LNP vaccine at 75 mcg weekly for the first 4 doses and a 5th dose 1 month after the 4th dose.
  Other Names: PD-1 mRNA LNP vaccine at 75 mcg
  Arms: Medium Dose
Drug: High dose PD-1 mRNA LNP vaccines — Patients will receive PD-1 mRNA LNP vaccine at 100 mcg weekly for the first 4 doses and a 5th dose 1 month after the 4th dose.
  Other Names: PD-1 mRNA LNP vaccine at 100 mcg
  Arms: High Dose

SUMMARY:
Evaluating the Safety and Efficacy of PD-1 mRNA LNP Vaccine Therapy in Patients with Primary Hepatocellular Carcinoma Who Have Failed Advanced Standard Therapy

DETAILED DESCRIPTION:
PD-1 mRNA LNP is an immune checkpoint mRNA vaccine loaded with the gene coding for the PD-1 protein Safety, tolerability, immunogenicity and preliminary efficacy of mRNA vaccines with PD-1 as the immunogen in the treatment of primary liver cancer. The aim of this study is to establish a novel PD-1-based mRNA for the treatment of advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients: ≥18 years of age; ≤70 years of age;
2. Recurrent or metastatic hepatocellular carcinoma that has failed second-line standard therapy.
3. Patients with at least one target lesion with a measurable diameter according to the RECIST criteria (CT scan of tumor lesions with a long diameter of ≥10mm, CT scan of lymph node lesions with a short diameter of ≥10mm and a layer thickness of no more than 5mm);
4. ECOG physical condition score: 0 to 1;
5. Expected survival ≥ 3 months;
6. Good function of major organs, i.e., relevant examination indexes within 14 days prior to randomization meet the following requirements:

   * Routine blood tests: hemoglobin ≥80g/L (no blood transfusion within 14 days); neutrophil count >1.5×109 /L; platelet count ≥80×109 /L;
   * Biochemical tests: total bilirubin ≤1.5 × ULN (upper limit of normal); blood alanine aminotransferase (ALT) or blood alanine transaminase (AST) ≤ 2.5 × ULN; if liver metastases, ALT or AST ≤ 5 × ULN; endogenous creatinine clearance ≥ 60 ml/min (Cockcroft-Gault formula);
   * cardiac Doppler ultrasound: left ventricular ejection fraction (LVEF) (LVEF) ≥50%.
7. Good compliance and family agreement to cooperate in receiving survival follow-up.

Exclusion Criteria:

1. Participation in a clinical trial of another drug within 4 weeks;
2. Patients with a prior history of other neoplasms, unless cervical cancer in situ, treated squamous skin cancer or epithelial tumor of the bladder or other malignancies that have undergone radical therapy (at least 5 years prior to enrollment);
3. Patients with uncontrolled cardiac clinical symptoms or disease, such as NYHA class 2 or higher heart failure, unstable angina pectoris , myocardial infarction within 1 year, clinically significant Supraventricular or ventricular arrhythmias requiring treatment or intervention.
4. For female subjects: women who are pregnant or breastfeeding.
5. Patients with active tuberculosis, bacterial or fungal infection (≥ grade 2 of NCI-CTCAE 5.0); HIV infection; active HBV infection; HCV infection.
6. Those with a history of psychotropic substance abuse that they are unable to abstain from or those with mental disorders;
7. Subjects with any active autoimmune disease or history of autoimmune disease (e.g., the following, but not limited to : uveitis, enteritis, pituitary gland inflammation, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or asthma that has resolved completely in childhood and does not require any intervention in adulthood may be enrolled; subjects with asthma requiring medical intervention with bronchodilators may not be enrolled).
8. Patients who have been inoculated with mRNA drugs.
9. Participation in clinical trials involving lipid nanoparticles, a component of the study vaccine.
10. Contraindications to intramuscular injection.
11. History of substance abuse or known medical, psychological or social conditions such as alcohol or drug abuse.
12. Known allergy, hypersensitivity or intolerance to the investigational vaccine (including any excipients). Previous history of severe allergy to any drug, food, or vaccination, such as anaphylaxis, allergic laryngeal edema, allergic dyspnea, anaphylactic purpura, thrombocytopenic purpura, localized anaphylactic necrotic reaction (Arthus reaction).
13. The female subject is planning to become pregnant or the male subject's partner is planning to become pregnant during the Screening Period and up to 12 months after the full course of drug administration.
14. In the judgment of the investigator, there is a serious concomitant disease that jeopardizes the patient's safety or interferes with the patient's ability to complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  The ratio of participants assessed with complete response (CR) or partial response(PR) as a best overall response.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 2 years
  The ratio of subjects assessed with CR or PR or stable disease (SD) as a best overalresponse.
DRR (Durable Response Rate) | 2 years
  DRR is defined as the proportion of objective response (CR and PR as determined by the investigator) lasting at least 6 months at any time within 12 months of initiation of treatment.
DOR (Duration of Response) | 2 years
  DOR is defined as the time from the date when the PR is first recorded or better to the date when the disease progression is first recorded (for the responder, i.e., PR or better). Responders who did not record disease progress will be censored on the date that the last assessment was SD or better.
TTR (Response Time） | 2 years
  TTR is defined as the time from the date of the first administration to the date of the first record of the objective tumor response (CR and PR determined by the investigator).
PFS (progression-free survival) | 2 years
  PFS is defined as the duration until disease progression or death in participants fromthe first dose of immunization.
OS (Overall Survival) | 2 years
  0S is defined as the duration until death in participants from the first dose ofimmunization.
TTP (Time to Progression) | 2 years
  TTP is defined as the time from the date of first dose to the date of first documented disease progression, as defined by standard disease criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — West China Hospital
Locations (2):
- China (2):
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan University West China Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen X, Wu Y, Yang T, Wei M, Wang Y, Deng X, Shen C, Li W, Zhang H, Xu W, Gou L, Zeng Y, Zhang Y, Wang Z, Yang J. Salidroside alleviates cachexia symptoms in mouse models of cancer cachexia via activating mTOR signalling. J Cachexia Sarcopenia Muscle. 2016 May;7(2):225-32. doi: 10.1002/jcsm.12054. Epub 2016 Jan 18. PMID 27493875
- [Result] Wu Y, Li W, Chen X, Wang H, Su S, Xu Y, Deng X, Yang T, Wei M, Li L, Liu Y, Yang J, Li W. DOG1 as a novel antibody-drug conjugate target for the treatment of multiple gastrointestinal tumors and liver metastasis. Front Immunol. 2023 Jan 26;14:1051506. doi: 10.3389/fimmu.2023.1051506. eCollection 2023. PMID 36776873
- [Result] Sabnis S, Kumarasinghe ES, Salerno T, Mihai C, Ketova T, Senn JJ, Lynn A, Bulychev A, McFadyen I, Chan J, Almarsson O, Stanton MG, Benenato KE. A Novel Amino Lipid Series for mRNA Delivery: Improved Endosomal Escape and Sustained Pharmacology and Safety in Non-human Primates. Mol Ther. 2018 Jun 6;26(6):1509-1519. doi: 10.1016/j.ymthe.2018.03.010. Epub 2018 Mar 14. PMID 29653760
- [Result] Selvaggio G, Leonardelli L, Lofano G, Fresnay S, Parolo S, Medini D, Siena E, Marchetti L. A quantitative systems pharmacology approach to support mRNA vaccine development and optimization. CPT Pharmacometrics Syst Pharmacol. 2021 Dec;10(12):1448-1451. doi: 10.1002/psp4.12721. Epub 2021 Oct 21. No abstract available. PMID 34672423
- [Result] Xu S, Yang K, Li R, Zhang L. mRNA Vaccine Era-Mechanisms, Drug Platform and Clinical Prospection. Int J Mol Sci. 2020 Sep 9;21(18):6582. doi: 10.3390/ijms21186582. PMID 32916818
- [Result] Linares-Fernandez S, Lacroix C, Exposito JY, Verrier B. Tailoring mRNA Vaccine to Balance Innate/Adaptive Immune Response. Trends Mol Med. 2020 Mar;26(3):311-323. doi: 10.1016/j.molmed.2019.10.002. Epub 2019 Nov 5. PMID 31699497
- [Result] Verbeke R, Hogan MJ, Lore K, Pardi N. Innate immune mechanisms of mRNA vaccines. Immunity. 2022 Nov 8;55(11):1993-2005. doi: 10.1016/j.immuni.2022.10.014. PMID 36351374
- [Result] Lim SA, Cox A, Tung M, Chung EJ. Clinical progress of nanomedicine-based RNA therapies. Bioact Mater. 2021 Oct 22;12:203-213. doi: 10.1016/j.bioactmat.2021.10.018. eCollection 2022 Jun. PMID 35310381
- [Result] Sebastian M, Schroder A, Scheel B, Hong HS, Muth A, von Boehmer L, Zippelius A, Mayer F, Reck M, Atanackovic D, Thomas M, Schneller F, Stohlmacher J, Bernhard H, Groschel A, Lander T, Probst J, Strack T, Wiegand V, Gnad-Vogt U, Kallen KJ, Hoerr I, von der Muelbe F, Fotin-Mleczek M, Knuth A, Koch SD. A phase I/IIa study of the mRNA-based cancer immunotherapy CV9201 in patients with stage IIIB/IV non-small cell lung cancer. Cancer Immunol Immunother. 2019 May;68(5):799-812. doi: 10.1007/s00262-019-02315-x. Epub 2019 Feb 15. PMID 30770959
- [Result] Hong HS, Koch SD, Scheel B, Gnad-Vogt U, Schroder A, Kallen KJ, Wiegand V, Backert L, Kohlbacher O, Hoerr I, Fotin-Mleczek M, Billingsley JM. Distinct transcriptional changes in non-small cell lung cancer patients associated with multi-antigenic RNActive(R) CV9201 immunotherapy. Oncoimmunology. 2016 Nov 18;5(12):e1249560. doi: 10.1080/2162402X.2016.1249560. eCollection 2016. PMID 28123889
- [Result] Lorentzen CL, Haanen JB, Met O, Svane IM. Clinical advances and ongoing trials on mRNA vaccines for cancer treatment. Lancet Oncol. 2022 Oct;23(10):e450-e458. doi: 10.1016/S1470-2045(22)00372-2. PMID 36174631
- [Result] Yuan Y, Gao F, Chang Y, Zhao Q, He X. Advances of mRNA vaccine in tumor: a maze of opportunities and challenges. Biomark Res. 2023 Jan 18;11(1):6. doi: 10.1186/s40364-023-00449-w. PMID 36650562
- [Result] Miao L, Zhang Y, Huang L. mRNA vaccine for cancer immunotherapy. Mol Cancer. 2021 Feb 25;20(1):41. doi: 10.1186/s12943-021-01335-5. PMID 33632261